CLINICAL TRIAL: NCT05730010
Title: Discerning the Impact of ctDNA Detection on Patient Decision Making in Early Stage Breast Cancer: a Conjoint Analysis
Status: Completed | Type: Observational
Sponsor: Indiana University (Other)
Responsible Party: Principal Investigator, Tarah J Ballinger, MD, Assistant Professor of Clinical Medicine, Indiana University
Other Study IDs: CTO-IUSCCC-0803
Record Dates: First submitted 2023-01-31; First posted 2023-02-15 (Actual); Last update posted 2023-08-03 (Actual); Status verified 2023-08

CONDITIONS: Triple Negative Breast Cancer
Keywords: breast cancer, ctDNA
MeSH Terms: conditions — Triple Negative Breast Neoplasms; Breast Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study will examine how ctDNA and additional prognostic genomic information in patients with early stage breast cancer might influences patient decision- making regarding systemic therapy options.

DETAILED DESCRIPTION:
This study is an electronically delivered, one time cross sectional survey study. The investigators want to understand how patients with triple negative breast cancer at high risk for disease recurrence will prioritize additional benefit over toxicity when considering treatment options, and if their knowledge of ctDNA positivity versus negativity will further shift this balance toward benefit.

ELIGIBILITY:
Inclusion Criteria:

* Self- reported history of non-metastatic breast cancer
* Self- reported history of receiving chemotherapy for breast cancer
* Self- reported history of chemotherapy completed at least 6 months ago but no more than 10 years ago
* Able to complete an online survey
* English speaking

Exclusion Criteria:

N/A

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Approximately 200 subjects will be recruited by Research Advocacy Network (RAN) and their partner organizations through email and social media solicitation.
Sampling Method: Probability Sample
Enrollment: 289 (Actual)
Dates: Start 2023-04-16 (Actual); Primary Completion 2023-06-26 (Actual); Study Completion 2023-06-26 (Actual)

PRIMARY OUTCOMES:
Examine whether knowledge of ctDNA negativity influences patient decision-making | Once all surveys in the sample size are completed, 6 months anticipated
  Ratings- based analysis will be used to examine whether knowledge of ctDNA negativity increases patient acceptability (and if so, by how much) of no therapy in the adjuvant setting, compared to standard of care capecitabine.

SECONDARY OUTCOMES:
Estimate at what degree of benefit a given treatment would be acceptable to patients | Once all surveys in the sample size are completed, 6 months anticipated
  When assuming risk of recurrence of ctDNA positivity, we will use ratings- based conjoint analysis to determine part-worth utilities of each attribute - potential toxicity and potential benefit. Comparison of part-worth utilities will be used to estimate at what degree of benefit a given treatment would be acceptable, which will inform future trials.

CONTACTS AND LOCATIONS:
Locations (1):
- Indiana University Melvin and Bren Simon Comprehensive Cancer Center, Indianapolis, Indiana, United States